CLINICAL TRIAL: NCT06238232
Title: 68Ga-Pentixafor PET/CT Versus Adrenal Vein Sampling to Determine Treatment in Primary Aldosteronism: A Multicenter Randomized Clinical Trial
Brief Title: Outcome of 68Ga-Pentixafor PET/CT Versus Adrenal Vein Sampling in Primary Aldosteronism
Acronym: GAPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qifu Li (Other)
Collaborators: The Affiliated Hospital Of Southwest Medical University (Other); West China Hospital (Other); Tongji Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The Third Xiangya Hospital of Central South University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Changzhi Medical College (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor-Investigator, Qifu Li, Primary investigator, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: GAPA study
Record Dates: First submitted 2024-01-04; First posted 2024-02-02 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Primary Aldosteronism
Keywords: Primary aldosteronism;; Adrenal venous sampling; 68Ga-Pentixafor PET/CT; outcome; multicenter randomized
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 68Ga-Pentixafor PET/CT group (Experimental): Patients divided into 68Ga-Pentixafor PET/CT group need to undergo 68Ga-Pentixafor PET/CT examination and guide subsequent treatment based on the results
  Interventions: Diagnostic Test: 68Ga-Pentixafor PET/CT
- AVS group (No Intervention): Patients divided into AVS group need to undergo AVS to guide subsequent treatment based on the results

INTERVENTIONS:
Diagnostic Test: 68Ga-Pentixafor PET/CT — The patients had a normal diet with no special preparation before 68Ga-Pentixafor PET/CT imaging. The dosage of intravenously injected 68Ga-Pentixafor was calculated based on the patient's weight (1.85 MBq [0.05mCi]/kg). Local PET/CT scanning of the upper abdomen was performed on a hybrid PET/CT scanner at 10 minutes after the injection of the intravenous tracer, respectively.
  Arms: 68Ga-Pentixafor PET/CT group

SUMMARY:
To compare the 68Ga-Pentixafor PET/CT and adrenal vein sampling on the long-term outcomes of primary aldosteronism (PA) patients with adrenal nodule (≥1cm)

DETAILED DESCRIPTION:
This is a randomized study involving patients with primary aldosteronism (PA) patients with adrenal nodule (≥1cm) who completed AVS or 68Ga-Pentixafor PET/CT.We will enroll 320 PA patients with adrenal nodule (≥1cm) .All paticipants will be randomized into 68Ga-Pentixafor PET/CT group(Intervention group) and AVS group(Control group) to compare the long-term outcomes of patients with PA.

ELIGIBILITY:
Inclusion Criteria:

(1)Getting the written informed consent (2)ARR ≥20 (pg/ml)/ (μIU/ml) or ARR ≥ 30(ng/dL)/(ng/ml/hr) plus at least one positive PA confirmatory test (CCT, SSIT).

(3)Patients who are willing to undergo surgery. (4)Patients with hypertension aged 18-70 years. (5)CT or MRI scan of the adrenal glands with nodule (≥1cm). Exclusion criteria

1. Combined with autonomous cortisol secretion, cortisol after 1mg dexamethasone suppression test (DST) ≥50 nmol/l.
2. PA patients who meet the by-passing AVS criteria [i.e., younger than 35 years old, spontaneous hypokalemia, adrenal CT indicated unilateral low-density adenoma (≥1cm), plasma aldosterone >300pg/ml]
3. Suspicion of familial hyperaldosteronism or Liddle syndrome. [i.e., age <20 years, hypertension and hypokalemia, or with family history]
4. Suspicion of pheochromocytoma or adrenal carcinoma.
5. Patients with actively malignant tumor.
6. Patients who have adrenalectomy history or with adrenocortical insufficiency.
7. Long-term use of glucocorticoids.
8. Pregnant or lactating women; with alcohol or drug abuse and mental disorders.
9. Congestive heart failure with New York Heart Association (NYHA) Functional Classification III or IV; History of serious cardiovascular or cerebrovascular disease (angina, myocardial infarction or stroke) in the past 3 months; Severe anemia (Hb<60g/L); Serious liver dysfunction or chronic kidney disease aspartate aminotransferase (AST) or alanine transaminase (ALT) >3 times the upper limit of normal, or estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73 m2); Systemic Inflammatory Response Syndrome (SIRS); Uncontrolled diabetes (FBG≥13.3 mmol/L); Obesity (BMI≥35 kg/m²) or Underweight (BMI≤18 kg/m²); Untreated aneurysm; Other comorbidity potentially interfering with treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of complete biochemical remission | At 6 months of follow-up.
  Blood was drawn to measure aldosterone, renin and potassium.According to PASO criteria, outcomes of adrenalectomy for unilateral primary aldosteronism were classified into complete, partial, and absent success, for both clinical and biochemical outcomes.The proportion of complete biochemical remission according to PASO consensus criteria.

SECONDARY OUTCOMES:
The proportion of complete clinical remission | At 6 months of follow-up.
  Blood was drawn to measure aldosterone, renin and potassium.According to PASO criteria, outcomes of adrenalectomy for unilateral primary aldosteronism were classified into complete, partial, and absent success, for both clinical and biochemical outcomes.The proportion of complete biochemical remission according to PASO consensus criteria.
In surgical population, the proportion of complete biochemical remission | At 6 months of follow-up.
  Blood was drawn to measure aldosterone, renin and potassium.According to PASO criteria, outcomes of adrenalectomy for unilateral primary aldosteronism were classified into complete, partial, and absent success, for both clinical and biochemical outcomes.The proportion of complete biochemical remission according to PASO consensus criteria.
In surgical population, the proportion of complete clinical remission | At 6 months of follow-up.
  Blood was drawn to measure aldosterone, renin and potassium.According to PASO criteria, outcomes of adrenalectomy for unilateral primary aldosteronism were classified into complete, partial, and absent success, for both clinical and biochemical outcomes.The proportion of complete biochemical remission according to PASO consensus criteria.
Daily defined doses (DDD) of antihypertensive agents | At 6-12 months of follow-up.
  Prescribed daily dose (DDD) of antihypertensive drugs (including MRA) in each group after 6-12 months of follow-up.
Total cost of diagnosis and treatment | At baseline and 6 months of follow-up.
  After patients are determined to be enrolled, treatment costs incurred for the diagnostic process will be calculated for each subject. This includes CT,AVS or PET/CT, surgery, medications, etc.
Health Related Quality of Life | At baseline and 6 months of follow-up.
  The quality of life in our patients may be influenced in different ways.AVS is an invasive test, PET/CT does not require any preparation of the patient before the test. Questionnaires of QOL-BREF will be conducted by patients before treatment and at 6-12 months follow-up in each group.This will allow for a detailed analysis of the impact of the two strategies on the quality of life of the patients.
Comparison of adverse events | At baseline and 6 month of follow-up.
  The occurrence of adverse events was recorded, including PET/CT contrast agent allergy, adrenal vein hemorrhage and related adrenal insufficiency, hypertensive emergency, anaphylactic shock, venous thrombosis, pulmonary embolism, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Qifu Li, PhD, Study Chair — the Chongqing Primary Aldosteronism Study (CONPASS) Group
Locations (1):
- The First Affilated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rossi GP, Bernini G, Caliumi C, Desideri G, Fabris B, Ferri C, Ganzaroli C, Giacchetti G, Letizia C, Maccario M, Mallamaci F, Mannelli M, Mattarello MJ, Moretti A, Palumbo G, Parenti G, Porteri E, Semplicini A, Rizzoni D, Rossi E, Boscaro M, Pessina AC, Mantero F; PAPY Study Investigators. A prospective study of the prevalence of primary aldosteronism in 1,125 hypertensive patients. J Am Coll Cardiol. 2006 Dec 5;48(11):2293-300. doi: 10.1016/j.jacc.2006.07.059. Epub 2006 Nov 13. PMID 17161262
- [Result] Xu Z, Yang J, Hu J, Song Y, He W, Luo T, Cheng Q, Ma L, Luo R, Fuller PJ, Cai J, Li Q, Yang S; Chongqing Primary Aldosteronism Study (CONPASS) Group. Primary Aldosteronism in Patients in China With Recently Detected Hypertension. J Am Coll Cardiol. 2020 Apr 28;75(16):1913-1922. doi: 10.1016/j.jacc.2020.02.052. PMID 32327102
- [Result] Mulatero P, Sechi LA, Williams TA, Lenders JWM, Reincke M, Satoh F, Januszewicz A, Naruse M, Doumas M, Veglio F, Wu VC, Widimsky J. Subtype diagnosis, treatment, complications and outcomes of primary aldosteronism and future direction of research: a position statement and consensus of the Working Group on Endocrine Hypertension of the European Society of Hypertension. J Hypertens. 2020 Oct;38(10):1929-1936. doi: 10.1097/HJH.0000000000002520. PMID 32890265
- [Result] Monticone S, D'Ascenzo F, Moretti C, Williams TA, Veglio F, Gaita F, Mulatero P. Cardiovascular events and target organ damage in primary aldosteronism compared with essential hypertension: a systematic review and meta-analysis. Lancet Diabetes Endocrinol. 2018 Jan;6(1):41-50. doi: 10.1016/S2213-8587(17)30319-4. Epub 2017 Nov 9. PMID 29129575
- [Result] Hundemer GL, Curhan GC, Yozamp N, Wang M, Vaidya A. Renal Outcomes in Medically and Surgically Treated Primary Aldosteronism. Hypertension. 2018 Sep;72(3):658-666. doi: 10.1161/HYPERTENSIONAHA.118.11568. PMID 29987110
- [Result] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Result] Amar L, Baguet JP, Bardet S, Chaffanjon P, Chamontin B, Douillard C, Durieux P, Girerd X, Gosse P, Hernigou A, Herpin D, Houillier P, Jeunemaitre X, Joffre F, Kraimps JL, Lefebvre H, Menegaux F, Mounier-Vehier C, Nussberger J, Pagny JY, Pechere A, Plouin PF, Reznik Y, Steichen O, Tabarin A, Zennaro MC, Zinzindohoue F, Chabre O. SFE/SFHTA/AFCE primary aldosteronism consensus: Introduction and handbook. Ann Endocrinol (Paris). 2016 Jul;77(3):179-86. doi: 10.1016/j.ando.2016.05.001. Epub 2016 Jun 15. PMID 27315757
- [Result] Nishikawa T, Omura M, Satoh F, Shibata H, Takahashi K, Tamura N, Tanabe A; Task Force Committee on Primary Aldosteronism, The Japan Endocrine Society. Guidelines for the diagnosis and treatment of primary aldosteronism--the Japan Endocrine Society 2009. Endocr J. 2011;58(9):711-21. doi: 10.1507/endocrj.ej11-0133. Epub 2011 Aug 9. PMID 21828936
- [Result] Young WF, Stanson AW, Thompson GB, Grant CS, Farley DR, van Heerden JA. Role for adrenal venous sampling in primary aldosteronism. Surgery. 2004 Dec;136(6):1227-35. doi: 10.1016/j.surg.2004.06.051. PMID 15657580
- [Result] Scala S. Molecular Pathways: Targeting the CXCR4-CXCL12 Axis--Untapped Potential in the Tumor Microenvironment. Clin Cancer Res. 2015 Oct 1;21(19):4278-85. doi: 10.1158/1078-0432.CCR-14-0914. Epub 2015 Jul 21. PMID 26199389
- [Result] Heinze B, Fuss CT, Mulatero P, Beuschlein F, Reincke M, Mustafa M, Schirbel A, Deutschbein T, Williams TA, Rhayem Y, Quinkler M, Rayes N, Monticone S, Wild V, Gomez-Sanchez CE, Reis AC, Petersenn S, Wester HJ, Kropf S, Fassnacht M, Lang K, Herrmann K, Buck AK, Bluemel C, Hahner S. Targeting CXCR4 (CXC Chemokine Receptor Type 4) for Molecular Imaging of Aldosterone-Producing Adenoma. Hypertension. 2018 Feb;71(2):317-325. doi: 10.1161/HYPERTENSIONAHA.117.09975. Epub 2017 Dec 26. PMID 29279316
- [Result] Hu J, Xu T, Shen H, Song Y, Yang J, Zhang A, Ding H, Xing N, Li Z, Qiu L, Ma L, Yang Y, Feng Z, Du Z, He W, Sun Y, Cai J, Li Q, Chen Y, Yang S; Chongqing Primary Aldosteronism Study (CONPASS) Group. Accuracy of Gallium-68 Pentixafor Positron Emission Tomography-Computed Tomography for Subtyping Diagnosis of Primary Aldosteronism. JAMA Netw Open. 2023 Feb 1;6(2):e2255609. doi: 10.1001/jamanetworkopen.2022.55609. PMID 36795418
- [Result] Ding J, Zhang Y, Wen J, Zhang H, Wang H, Luo Y, Pan Q, Zhu W, Wang X, Yao S, Kreissl MC, Hacker M, Tong A, Huo L, Li X. Imaging CXCR4 expression in patients with suspected primary hyperaldosteronism. Eur J Nucl Med Mol Imaging. 2020 Oct;47(11):2656-2665. doi: 10.1007/s00259-020-04722-0. Epub 2020 Mar 23. PMID 32206838